CLINICAL TRIAL: NCT05325320
Title: Reducing Serious Mental Illness and Suicide Stigma Among Medical Students
Brief Title: Intervention to Reduce Serious Mental Illness and Suicide Stigma Among Medical Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34MH120179-01A1 (NIH); 1R34MH120179-01A1 (NIH)
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Stigmatization; Clinical Competence
MeSH Terms: conditions — Stereotyping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stigma Reduction Intervention (Experimental): Participants randomized to the experimental condition will receive the SMI/SIA Stigma Reduction Intervention.
  Interventions: Behavioral: SMI/SIA Stigma Reduction Intervention
- Disaster Preparedness Course (Other): Participants randomized to the control condition will receive a Disaster Preparedness Course, addressing the basics of natural disaster preparedness.
  Interventions: Other: Disaster Preparedness Course

INTERVENTIONS:
Behavioral: SMI/SIA Stigma Reduction Intervention — Online course designed to reduce stigma behaviors towards serious mental illness and suicide ideation and attempt among medical students. It aims to improve medical students' healthcare delivery skills.
  Arms: Stigma Reduction Intervention
Other: Disaster Preparedness Course — Online course designed to improve professionals' skills and competencies for engaging in disaster preparedness.
  Arms: Disaster Preparedness Course

SUMMARY:
The team aims to develop and test the efficacy of a serious mental illness (SMI) and suicide ideation and attempt (SIA) stigma reduction intervention for medical students. The team expects that after intervention exposure, relative to control group, participants in the experimental condition will manifest more favorable change in knowledge, attitudes, and behaviors.

DETAILED DESCRIPTION:
People with serious mental illness (PSMI; i.e. Schizophrenia and bipolar disorder) die, on average, 25 years earlier than the general population. Suicide is a key factor for this disparity as it is the leading cause of unnatural deaths among this population. Research identifies Latinos as a particularly vulnerable group, accounting for one of the highest rates (over 30%) of serious mental illness (SMI) among ethnic minorities in the United States (US). Latinos also hold one of the highest prevalence of suicide ideation and attempts (SIA) with rates of 10.1% and 4.4% respectively. This scenario worsens for one Latino subgroup, Puerto Ricans, who have the highest prevalence of SMI (36%) and SIA among Latinos in the US (7.9% and 3.5% respectively). Taken together, these facts present a concerning scenario for Latinos, especially Puerto Ricans with SMI/SIA. Health professionals play a key role in identifying SMI/SIA among patients; unfortunately, SMI/SIA stigma hinders this process.

The proposed study aims to: 1) develop the content of an intervention to reduce SMI/SIA stigma among medical students, 2) determine the acceptability and feasibility of implementing the intervention among medical students by examining recruitment/screening procedures, participation/refusal/retention rates, and participant satisfaction, and; 3) pilot test the preliminary efficacy of the intervention in reducing SMI/SIA stigma among medical students by increasing knowledge of SMI and SIA, reducing negative attitudes towards SMI/SIA and increasing behavioral skills for providing healthcare to PSMI.

ELIGIBILITY:
Inclusion Criteria:

* Medical student currently in third year of medical school training

Exclusion Criteria:

* Do not speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Increase from baseline in scores on the Behavioral Health Skills Inventory (BHSI) | Baseline, immediately after intervention, 2 week follow-up
  This 29-item inventory assesses standardized patient simulation interactions including three behavioral components addressing general healthcare related behaviors, SMI related behaviors and SIA related behaviors. Scores range from 0 to 58, with higher numbers reflecting higher skills in healthcare service delivery for PSMI/SIA.

SECONDARY OUTCOMES:
Increase from baseline in scores on the Serious Mental Illness Literacy Scale | Baseline, immediately after intervention, 2 week follow-up
  This adapted and pilot tested version of the Mental Health Literacy Scale, measures participants' knowledge regarding SMI. The Scale addresses the ability to recognize SMI including: Bipolar Disorder and Schizophrenia. The Scale is composed of two sections measuring SMI knowledge. The first is composed of 15 items (4-point Likert Scale) ranging from (1) very unlikely to (4) very likely. The second section is composed of 20 items using a 5-point Likert Scale ranging from (1) strongly disagree to (5) strongly agree.
Increase from baseline in scores on the Literacy of Suicide Scale (LOSS) | Baseline, immediately after intervention, 2 week follow-up
  This SIA knowledge measure is answered in a correct/incorrect/don't know format. The 27 items are rated on a 3-point scale (true, false, or I don't know), with correct responses allocated a score of 1 and incorrect or I don't know responses assigned a score of 0. Higher LOSS scores indicate higher suicide literacy.
Decrease from baseline in scores on The Mental Health Stigma Scale for Health Professionals | Baseline, immediately after intervention, 2 week follow-up
  Used to evaluate mental illness stigma among health professionals, including medical students. This 12-item measure uses a 5-point Likert from (1) strongly agree to (5) strongly disagree. It has three dimensions (social distance, negative character attributions, and self-sufficiency problems).
Decrease from Stigma of Suicide Scale (Short Version) | Baseline, immediately after intervention, 2 week follow-up
  This three-factor scale measures stigma towards people who die by suicide. This short version consists of 16-items. Each item consists of a one-word descriptor of a person who dies by suicide, rated on a 5-point Likert scale from (1) strongly disagree to (5) strongly agree.
Decrease from baseline in scores on The Emotional Reactions Scale | Baseline, immediately after intervention, 2 week follow-up
  This scale was adapted from the original Emotional Reactions to the Mentally Ill Scale to include a suicide ideation case. This 9-item scale includes two vignettes of a person with SIA to assess emotional reaction to the scenario. Each item is rated in a 5-point Likert scale.
Increase from baseline in scores on the Cross-Cultural Care Scale (CCCS) | Baseline, immediately after intervention, 2 week follow-up
  This adaptation of the Cross- Cultural Care Scale which assesses preparedness to treat diverse patient populations. This 19-item scale is rated in a 5-point Likert format.

OTHER OUTCOMES:
Intervention Contamination Inventory | Immediately after intervention, 2 week follow-up
  This inventory includes four closed- and open-ended questions addressing the following contamination-related areas: receiving information on SMI/SIA topics from another source, participation in other SMI/SIA courses or workshops, and type of information received in them. Via coding of both the closed and open-ended question contamination will be defined via yes-no variable (0 = no contamination reported; 1 = contamination reported).
Intervention Acceptability Questionnaire | Immediately after intervention, 2 week follow-up
  This questionnaire includes 16 items addressing participants' satisfaction with the intervention's format, content, and delivery. The study team has successfully used this questionnaire in intervention development studies and has adapted it for the proposed study.
Social Desirability Scale | Immediately after intervention, 2 week follow-up
  This scale is composed of 11 items rated on a 4-point Likert scale ranging from (1) "Strongly Disagree" to (4) "Strongly Agree". This measure has excellent reliability coefficients with Cronbach alphas of .86 when used with medical students.

CONTACTS AND LOCATIONS:
Overall Officials: Eliut Rivera-Segarra, Ph.D, Principal Investigator — Ponce Health Sciences University; Nelson Varas-Diaz, Ph.D, Principal Investigator — Florida International University
Locations (2):
- Florida International University, Miami, Florida, United States
- Ponce Health Sciences University, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No